CLINICAL TRIAL: NCT03775395
Title: Hepatic Artery Infusion Chemotherapy Plus Lenvatinib vs Hepatic Artery Infusion Chemotherapy Plus Sorafenib for Advanced Hepatocellular Carcinoma
Brief Title: HAIC Plus Lenvatinib vs HAIC Plus Sorafenib for Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCC-S055
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatic artery infusion chemotherapy; Sorafenib; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC plus Lenvatinib (Experimental)
  Interventions: Drug: Lenvatinib; Procedure: Hepatic arterial infusion chemotherapy
- HAIC plus Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib; Procedure: Hepatic arterial infusion chemotherapy

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Arms: HAIC plus Lenvatinib
Drug: Sorafenib — 400mg BID daily oral dosing
  Arms: HAIC plus Sorafenib
Procedure: Hepatic arterial infusion chemotherapy — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) compared with lenvatinib combined with HAIC in patients with advanced hepatocellular carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 30mmol/L
* Serum albumin ≥ 30 g/L
* ASL and AST ≤ 5 x upper limit of normal
* Serum creatinine ≤ 1.5 x upper limit of normal
* INR ≤ 1.5 or PT/APTT within normal limits
* Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time Frame: 12 months
  Overall survival

SECONDARY OUTCOMES:
Time to progression | Time Frame: 12 months
  Time to progression
Adverse Events | [Time Frame: 30 days]
Progression Free Survival (PFS) | Time Frame: 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China